CLINICAL TRIAL: NCT01946672
Title: Individualisation du Drainage Lymphatique Des Membres inférieurs Lors du Curage Pelvien Pour Cancer gynécologique
Brief Title: Lower-Limb Drainage Mapping in Pelvic Lymphadenectomy for Gynaecological Cancer
Acronym: SENTIJAMBE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P110903
Record Dates: First submitted 2013-09-17; First posted 2013-09-19 (Estimated); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Gynaecological Malignant Tumours With Indication of Pelvic Lymphadenectomy
Keywords: gynaecological malignancy; pelvic lymphadenectomy; lymphedema; sentinel node; reverse mapping
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- isotopic intraoperative detection (Experimental): Lower-limb drainage isotopic intraoperative detection
  Interventions: Procedure: Lower-limb drainage isotopic intraoperative detection

INTERVENTIONS:
Procedure: Lower-limb drainage isotopic intraoperative detection — A radiopharmaceutical is injected into both feet on the day before surgery. Pelvic lower-limb drainage nodes (LLDNs) are identified using preoperative SPECT-CT and intraoperative isotopic probe detection, and then electively removed before complete pelvic lymphadenectomy. LLDNs and pelvic lymphadenectomy specimens undergo separate histological analysis.

SUMMARY:
The purpose of this study is to evaluate the feasibility of an isotopic technique to identify, and to map the lower-limb drainage nodes during pelvic lymphadenectomy for gynaecological cancers. The diagnostic value of our mapping method will be assessed, and we will determine the incidence of lymhedema.

DETAILED DESCRIPTION:
Pelvic lymphadenectomy is associated with a significant risk of lower-limb lymphedema. In this study, we evaluate the feasibility of identifying the lower-limb drainage nodes (LLDNs) during pelvic lymphadenectomy for gynaecological cancers using an isotopic detection technique with a preoperative radiopharmaceutical injection into both feet Secondary objectives are to map lower-limb drainage, to assess the diagnostic value of our mapping technique, and to determine the incidence of lymphedema. LLDN mapping may allow the preservation of LLDNs, thereby decreasing the risk of lower-limb lymphedema and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years of age or older with indication of pelvic lymphadenectomy for gynaecological malignancy:

  * High risk endometrial cancer (stage IB type I grade 3, stage I type II, stage> IB) or with metastatic sentinel lymph node,
  * Early cervical cancer, or with metastatic sentinel lymph node,
  * Ovarian cancer.
* Must provide her signed and informed consent
* Beneficiary of a health insurance
* Having received a medical examination

Exclusion Criteria:

* Contraindication to pelvic lymphadenectomy
* Presence of lymphedema of the lower limbs
* Contraindication to radiomarkers (allergy or hypersensitivity to any component of the biomarker)
* Patient with dementia or altered mental status
* Pregnant or breast feeding patients
* Participation in any other clinical trial that could interfere with the study results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Lower-limb drainage intraoperative isotopic detection rate in patients with pelvic lymphadenectomy for gynaecological cancers. | day of surgery

SECONDARY OUTCOMES:
Anatomy of lower-limb drainage | day of surgery
Percentage of patients with metastatic lower limb sampling | 2 weeks after surgery
Follow-up of patients to identify complications, and namely lower-limb lymphedema. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie BATS, MD, PhD, Principal Investigator — assistance publique des hopitaux de paris
Locations (1):
- HEGP, Paris, Île-de-France Region, France